CLINICAL TRIAL: NCT06338293
Title: Using OFR Software to Observe the Effects of Inclisiran Combined With Statins on the Morphology and Vascular Function of Coronary Vulnerable Plaques
Brief Title: Effects of Inclisiran Combined With Statins on the Morphology of Coronary Vulnerable Plaques
Acronym: EItoCVP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20240123-02
Record Dates: First submitted 2024-02-26; First posted 2024-03-29 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inclisiran＋rosuvastatin group (Experimental): Inclisiran sodium＋rosuvastatin 20mg group: Rosuvastatin was given 20mg daily for one year, and Inclisiran was given three times in total. After the first injection, 284mg(1.5ml solution) was injected subcutaneously, the second injection was 3 months after the first injection, and the third injection was in the ninth month.
  Interventions: Drug: Inclisiran sodium; Drug: Rosuvastatin
- Rosuvastatin group (Placebo Comparator): Rosuvastatin group: Rosuvastatin 20mg daily for one year.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Inclisiran sodium — The patients in Inclisiran group were given drugs three times in total. The first needle was injected subcutaneously with 284mg(1.5ml solution) after entering the group, the second needle was injected three months later and the third needle was injected at the ninth month.
  Arms: Inclisiran＋rosuvastatin group
Drug: Rosuvastatin — Rosuvastatin

SUMMARY:
Effects of inclisiran + statins vs. statins on the morphology and vascular function of coronary vulnerable plaques, in order to provide a better treatment and more detailed imaging basis for the treatment of coronary vulnerable plaques.

DETAILED DESCRIPTION:
The identification and treatment of vulnerable coronary plaques is still the focus of coronary heart disease research in recent several years. There are many methods to identify vulnerable plaque, such as NIRS, IVUS, OCT, but these methods have their own advantages and disadvantages, and they can't give the characteristics of diseased plaque completely and clearly. Therefore, if you want to better identify, track and treat vulnerable plaques, you need the comprehensive judgment of multi-modal detection methods, such as the comprehensive data of NIRS, IVUS, OCT, but in this case, there will be more and more invasive operations for patients, and the operation cost is high and time-consuming. OFR analysis software can quickly analyze the morphological and functional parameters of diseased vascular plaques based on OCT data, overcome the shortcomings of poor penetration of OCT and inability to observe the overall lesion contour, and can immediately give the morphological and functional parameters of diseased plaques, combining the data results of OCT, IVUS and FFR multimodal detection methods.

Statins have the effect of inducing regression and transforming coronary plaques into stability, but there are also some problems in the process of statin treatment. For example, for some patients with coronary heart disease, even the maximum tolerated dose of statins can not achieve the target goal of LDL-Cl; The side effects of statins, such as liver damage, muscle pain and blood sugar fluctuation, reduce the compliance of some patients. In recent years, the lipid-lowering effect of non-statins and the effect of stabilizing and reversing plaques have also attracted much attention, especially PCSK9 monoclonal antibody, such as, GLAGOV study, HUYGENS study, ALTAIR study and PACMAN-AMI study, compared with statins, they can reduce the plaques volume and stabilize the plaques morphology.

Inclisiran is the first siRNA drug in cardiovascular field. As a new generation of drugs acting on PCSK9, the current clinical research (ORION research series 1, 3, 8, 9, 10, 11) shows good lipid-lowering efficacy and safety tolerance. On the basis of statin therapy, LDL-C46%-55% is further reduced, which is more durable than monoclonal antibody, and the drug effect can last for half a year once used, and it has good safety and tolerance (except for the slight reaction of injection, there are almost no other side effects). So far, the research of Inclisiran mainly focuses on the safety and efficacy of lipid-lowering and the observation of clinical events, and the research on vulnerable plaque is very scarce. In this study, OFR analysis software will be used to observe whether Inclisiran combined with statin is superior to statin standard treatment on the vulnerable plaques, and it is expected to provide more superior clinical treatment scheme and more accurate imaging basis for identifying and treating vulnerable coronary plaques.

ELIGIBILITY:
Inclusion criteria: 1. Age 18-80 years old; 2. Coronary angiography (CAG) showed that the diameter of the primary coronary lesion was 20 ~ 70%, and the lesion was confirmed by OCT and OFR analysis, in which the target lesion contained at least one vulnerable plaque (the thinnest fibrous cap thickness was ≤65um, and the lipid core was ≥ 90), and the target vessel did not need further percutaneous coronary intervention (PCI); 3. Patients have been treated with statins for ≥4 weeks, but their LDL-C level were still ≥ 70 mg/dl (≥ 1.8 mmol/l).

Exclusion criteria: 1. Acute myocardial infarction occurred in recent 30 days; 2. The target lesion of coronary artery is severely distorted and angulated; Severe left main artery lesion, chronic occlusive lesion and bifurcation lesion; 3. Previous CABG; 4. Serum triglyceride (TG) > 500 mg/dl (> 5.6 mmol/l); 5. Patients with severe heart failure (< 40%) and respiratory failure; 6. Severe renal insufficiency (eGFR < 30ml ／min／1.73m2), active liver disease or severe liver damage;7. allergic to statins or inclisiran, and used PCSK9 monoclonal antibody in the past; 8. Known active infection or severe blood, metabolic or endocrine dysfunction; 9. Non-cardiac surgery is planned within 12 months; 10, can't follow the requirements of the follow-up, or researchers believe that the subjects to participate in the trial will increase the risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change rate of the thinnest fibrous cap of vulnerable plaque at the target vascular lesion from baseline to one-year follow-up(△ FCT%) | one-year
  The change rate of the thinnest fibrous cap of vulnerable plaque at the target vascular lesion from baseline to one-year follow-up(△ FCT%)

SECONDARY OUTCOMES:
The change rate of TAV and plaque load of the target vascular lesion; | one-year
  The change rate of TAV and plaque load of the target vascular lesion from baseline to one-year follow-up;
The change rate of lipid composition of plaque: including the lipid volume , the maximum area and angle of lipid, the length of vulnerable plaque, etc. | one-year
  The change rate of lipid composition of plaque: including the lipid volume from baseline to one-year follow-up , the maximum area and angle of lipid from baseline to one-year follow-up, the length of vulnerable plaque from baseline to one-year follow-up, etc.
The change rates of other components of plaque (fiber, calcification, crystal, macrophage) | one-year
  The change rates of other components of plaque from baseline to one-year follow-up (fiber, calcification, crystal, macrophage)
The change rates of lesion OFR and target vessel OFR | one-year
  The change rates of lesion OFR and target vessel OFR from baseline to one-year follow-up
The change rates of other indexes (low density lipoprotein level, Lp-PLA2, hs-CRP, etc.) | one-year
  The change rates of other indexes from baseline to one-year follow-up(low density lipoprotein level, Lp-PLA2, hs-CRP, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: China Jiangsu, Principal Investigator — Nanjin First Hospital,Nanjing Medical University
Locations (1):
- NanJing Frist Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No